CLINICAL TRIAL: NCT05056428
Title: Effects of Mindfulness Training on Emotional Care Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Lam Shui-fong, Director, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: UHongKong (JC PandA)
Record Dates: First submitted 2021-09-08; First posted 2021-09-24 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Mental Health Issue
Keywords: mindfulness; teacher mental health; emotional care; decentering; cognitive reappraisal; mindfulness-based intervention for teachers

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): 8-week mindfulness program
  Interventions: Behavioral: 8-week mindfulness program
- Wait-list control (No Intervention): Participants in wait-list control group will receive the same intervention, two months after experimental group completed the intervention.

INTERVENTIONS:
Behavioral: 8-week mindfulness program — The .b Foundations course is an 8-week mindfulness program developed by Mindfulness in Schools Project (MiSP) for school teachers and personnel. It includes a taster session and 8 weekly sessions. Each session lasts for 1.5 hours with a specific theme (e.g. Lesson 1 waking up from autopilot). Formal and informal mindfulness practices (e.g. mindful eating, body scan, mindful walking, habit releaser etc.), psychoeducation, cognitive exercises, inquiry, and home practice are involved.
  Arms: Intervention group

SUMMARY:
Teachers in Hong Kong are susceptible to professional stress and its associated psychosomatic illnesses. To enhance teachers' well-being, mindfulness training is conducted in local schools. The present study is a randomized controlled trial to investigate 1) the effects of mindfulness training on teachers' well-being (i.e. general health, positive affect, stress, negative affect); 2) whether decentering strategy (vs. cognitive reappraisal strategy) is nurtured by mindfulness practice; and 3) whether decentering instead of cognitive reappraisal is the mediator that explains the impact of mindfulness on well-being. Participants will be randomized to either intervention (8-week .b Foundations course) or waiting-list control condition.

DETAILED DESCRIPTION:
All the participants will complete an online survey before (baseline), after (post-intervention), and two-months (follow-up) after the intervention. A subset of participants (N = 30) will complete an electroencephalography (EEG) experiment.

Prior to the experiment, participants will complete an online questionnaire writing down eight recent autobiographical situations: four reflecting a neutral experience, two reflecting events that triggered anxiety, and two reflecting events that triggered sadness. After writing about each situation, participants will be asked to identify five keywords that are both unique and tightly linked to each situation.

During the experiment, participants will be reminded of the autobiographical situations in the computerized task. Participants will be asked to view the keywords (i.e. control condition); step back and view the keywords like an impartial observer, allowing whatever thoughts or emotions arise to come and go (i.e. decentering condition); and think about the keywords from different perspective to minimize negative emotions (i.e. reappraisal condition). EEG will be recorded while participants complete the task. Participants will receive $200 Hong Kong dollars each time as a remuneration for the time to participate in the experiment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years old or above
* Working in local schools or education institutions
* Willing to participate in mindfulness training voluntarily

Exclusion Criteria:

* Have history of neurological or psychiatric disorder, brain injury, birth complications, or significant sensory impairment
* Currently under medications that are known to affect the brain (e.g. anti-depressants, epileptica, tranquilizer, sleep medication, psychotropics, ritalin, concerta, etc.)
* Experiencing severe or unstable mental health condition currently
* Completed 8-week mindfulness training previously
* Unwilling to go by random assignment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2021-09-25 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Change in General Health | Baseline, Immediately after intervention, Two-months after intervention
  General Health Questionnaire (GHQ), 12 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Stress | Baseline, Immediately after intervention, Two-months after intervention
  Perceived Stress Scale (PSS), 10 items, 5-point Likert scale ranging from 1 (never) to 5 (always)

SECONDARY OUTCOMES:
Change in Positive affect | Baseline, Immediately after intervention, Two-months after intervention
  Positive and Negative Affect Schedule (PANAS), 4 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Negative affect | Baseline, Immediately after intervention, Two-months after intervention
  Positive and Negative Affect Schedule (PANAS), 4 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Decentering | Baseline, Immediately after intervention, Two-months after intervention
  Non Reactivity Subscale of Chinese Five Facet Mindfulness Questionnaire (FFMQ-C), 4 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Reappraisal | Baseline, Immediately after intervention, Two-months after intervention
  Reappraisal subscale of Emotion Regulation Questionnaire (ERQ), 6 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Mindfulness | Baseline, Immediately after intervention, Two-months after intervention
  Cognitive and Affective Mindfulness Scale-Revised (CAMS-R), 12 items, 5-point Likert scale ranging from 1 (never) to 5 (always)
Change in Late positive potential (LPP) | Baseline, Immediately after intervention
  A measure of emotional reactivity in EEG experiment; the amplitude of event-related potential (ERP) time-locked to the presentation of emotional stimulus (-200ms to 6000ms).

CONTACTS AND LOCATIONS:
Locations (1):
- Jockey Club "Peace and Awareness" Mindfulness Culture in Schools Initiative, Faculty of Social Sciences, The University of Hong Kong, Hong Kong, Hong Kong